CLINICAL TRIAL: NCT01182766
Title: High and Low Dose Topiramate for the Treatment of Alcohol-Dependent Smokers
Brief Title: New Treatment for Alcohol and Nicotine Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); M.D. Anderson Cancer Center (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Addiction Research and Education, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15597; 5R01AA019720-02 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-17 (Estimated); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Dependence; Nicotine Dependence
Keywords: alcohol; alcoholism; nicotine; cigarette
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder | interventions — Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-Dose Topiramate (Experimental): Low-dose topiramate (125 mg) with brief behavioral enhancement therapy
  Interventions: Drug: Low-Dose Topiramate
- High-Dose Topiramate (Experimental): High-dose topiramate (250 mg) with brief behavioral enhancement therapy
  Interventions: Drug: High-Dose Topiramate
- Placebo (Placebo Comparator): Placebo with brief behavioral enhancement therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-Dose Topiramate — Low-dose topiramate (up to 125 mg/day) with brief behavioral enhancement therapy
  Other Names: Topamax
  Arms: Low-Dose Topiramate
Drug: Placebo — Placebo with brief behavioral enhancement therapy
  Other Names: sugar pill
  Arms: Placebo
Drug: High-Dose Topiramate — High-dose topiramate (up to 250 mg/day) with brief behavioral enhancement therapy
  Other Names: Topamax
  Arms: High-Dose Topiramate

SUMMARY:
This research study aims to test whether topiramate (a drug that is being used for seizure) will help individuals who have problems with both alcohol and nicotine. The investigators believe that individuals taking topiramate will be more successful at abstaining from both alcohol and nicotine than individuals taking placebo.

DETAILED DESCRIPTION:
We propose a novel pharmacological strategy for treating alcohol and nicotine dependence concomitantly.

The reinforcing effects of both alcohol and nicotine are mediated through the cortico-mesolimbic dopamine (CMDA) system, and the concomitant use of both drugs enhances their pharmacological effects. We propose a better approach to control dopamine (DA) effects by contemporaneous indirect modulation of DA release and its functional expression. Both DA release from its cell bodies in the ventral tegmental area and the expression of its reinforcing effects through the cortico-mesolimbic system are modulated by gamma-aminobutyric acid (GABA) efferents under the tonic control of glutamate-mediated excitatory amino acid pathways. Thus, it is reasonable to hypothesize that a medication that facilitates cortico-mesolimbic GABAergic function and inhibits glutamate action should diminish both nicotine's and alcohol's reinforcing effects by inhibiting the release of midbrain DA and its functional expression through pathways projecting from the nucleus accumbens to the cortex. The promise of this novel approach is exemplified by our recent proof-of-concept demonstration that topiramate compared with placebo significantly improved smoking abstinence rates and decreased serum cotinine levels among alcohol dependent smokers. An important clinical effect of topiramate in alcohol-dependent individuals appears to be that its anti-withdrawal effects promote the gradual tapering of drinking. Hence, due to this unique anti-withdrawal effect of topiramate, we propose to adopt the same methodology for treating alcohol-dependent individuals, as is common practice with smokers, of setting a target quit date (TQD) after which relapse to either drug can be measured. We propose an 18-week, double-blind clinical trial with follow-up visits at 1 month and 3 months, in which alcohol-dependent smokers will receive brief behavioral compliance enhancement treatment (BBCET) plus a smoking self-help manual as their psychosocial treatment, and will be randomized to receive placebo,high-dose topiramate (up to 250 mg/day), or low-dose topiramate (up to 125 mg/day) to prevent relapse to heavy drinking and smoking. Each of the 3 treatment arms shall contain 98 individuals, with a total N of 294.

The TQD will occur at the beginning of the 6th week of treatment. Our primary objective is to determine whether both low- and high-dose topiramate will be more efficacious than placebo at reducing the percentage of heavy drinking days and increasing the continuous abstinence rate for smoking determined by a combination of self-report and carbon monoxide (CO) monitoring after the TQD and in the last 4 weeks of treatment. We also will be able to determine whether a lower dose of topiramate is as efficacious as the higher dose and, therefore, is associated with a lower adverse profile. Our secondary objectives are to test whether topiramate will be more efficacious than placebo at improving quality of life and reducing craving after the TQD and in the last 4 weeks of treatment and whether this improvement will be sustained in the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* Subjects must be above the age of 18
* Good physical health
* Diagnostic and Statistical Manual (DSM)-IV diagnosis of mild to severe alcohol use disorder
* Smoking ≥ 5 cigarettes/day
* Currently drinking at least 8 standard drink units (SDUs) per week for women and at least 15 SDUs per week in the 30 days prior to randomization
* Subjects must provide evidence of stable residence
* The pregnancy test for females of child-bearing potential at screen and prior to randomization must be negative. Additionally, women of child-bearing potential must be using an acceptable form of contraception.
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments
* Willing to participate in a treatment program for alcohol and nicotine dependence

Exclusion Criteria:

Please contact site for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, MD, Principal Investigator — University of Virginia; Robert M Anthenelli, MD, Principal Investigator — University of California, San Diego; Paul M Cinciripini, PHD, Principal Investigator — M.D. Anderson Cancer Center; Bankole A Johnson, MD, Principal Investigator — University of Virginia
Locations (4):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Center for Addiction Research & Education, Charlottesville, Virginia
  - University of Virginia Center for Addiction Research & Education, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: (UVA CARE Website) — https://med.virginia.edu/uva-clear/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 236 adults who met the DSM-5 criteria for Alcohol Use Disorder and Tobacco Use Disorder and recruited from three metropolitan areas in the U.S., including San Diego, California, Houston, Texas, and Charlottesville, Virginia. A Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnosis of mild to severe alcohol use disorder was required and participants must have smoked an average of 5 or more cigarettes/day in the 30 days prior to randomization.
Pre-assignment Details: Of 646 individuals who screened, 410 were excluded or uninterested. A total of 236 participants were enrolled and randomized into one of three study arms. Randomization was achieved using a block randomization procedure in which treatment groups were stratified to achieve a balance on age of onset for alcoholism (less than 26 years old or 26 years and older), gender, and drinks per drinking day (DDD) (< 8 DDD or ≥ 8 DDD) and the number of cigarettes smoked (<20 or >20 cigarettes/day).
Groups:
- Placebo: Participants received the 18-week placebo treatment with brief behavioral enhancement therapy
- Low-Dose Topiramate: Participants received the 18-week low-dose topiramate treatment (up to 125 mg/day) with brief behavioral enhancement therapy
- High-Dose Topiramate: Participants received the 18-week high-dose topiramate treatment (up to 250 mg/day) with brief behavioral enhancement therapy
Period: Overall Study
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
Started | 84 | 75 | 77
Completed | 36 | 35 | 41
Not Completed | 48 | 40 | 36
Not completed — Lost to Follow-up | 32 | 36 | 29
Not completed — Withdrawal by Subject | 14 | 3 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Non-compliance | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate | Total
Number analyzed (Participants) | 84 | 75 | 77 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.68 (10.35) | 48.07 (10.34) | 48.77 (9.86) | 48.16 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 25 | 76
  Male | 56 | 52 | 52 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 3 | 13
  Not Hispanic or Latino | 76 | 67 | 70 | 213
  Unknown or Not Reported | 3 | 3 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 29 | 31 | 22 | 82
  White | 46 | 36 | 48 | 130
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 6 | 22
Employment [Count of Participants; unit: Participants]
  Employed or student | 46 | 42 | 55 | 143
  Unemployed or retired | 36 | 28 | 18 | 82
  Employment unknown | 2 | 5 | 4 | 11
Baseline Smoking (CPD) [Mean (Standard Deviation); unit: cigarettes per day] | 21.34 (9.96) | 19.18 (10.47) | 20.33 (10.02) | 20.32 (10.14)
Baseline Drinking (SDU)/day [Mean (Standard Deviation); unit: standard drink units/day] | 10.02 (6.76) | 9.84 (5.51) | 9.88 (5.96) | 9.92 (6.10)
Mean Fagerström Test for Cigarette Dependence (FTCD) Score [Mean (Standard Deviation); unit: scores on a scale] — The Fagerstrom Test for Cigarette Dependence is a 6-question self-report scale used to assess nicotine dependence.The FTND score ranges from 0 to 10, with higher scores indicating greater dependence. Points from each question are summed together for a final score.
  0-2: Very low dependence 3-4: Low dependence 5: Medium dependence 6-7: High dependence 8-10: Very high dependence
  scores on a scale | 5.32 (1.92) | 5.27 (2.38) | 5.69 (2.30) | 5.42 (2.21)
AUDIT [Mean (Standard Deviation); unit: scores on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item questionnaire used to screen for hazardous and harmful alcohol consumption. It works by assessing alcohol consumption, drinking behavior, and alcohol-related problems. The total score ranges from 0 to 40, with higher scores more suggestive of alcohol use disorder.
  0 to 7 points: Low risk 8 to 15 points: Medium risk 16 to 19 points: High risk 20 to 40 points: Addiction likely
  scores on a scale | 21.39 (7.61) | 21.43 (7.23) | 19.40 (6.18) | 20.75 (7.08)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Smoking Abstinence in the Last 4 Weeks of Treatment Continuous Smoking Abstinence in the Last 4 Weeks of Treatment
Description: No smoking in the last 4 weeks of the 18-week treatment with an expired carbon monoxide level of <10 ppm as the biochemical verification. We used the intent-to-treat assumption, where missing smoking data were considered as smoking.
Time Frame: Week 15 - 18 of the 18-week medication treatment
Measure: Number; unit: participants
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
Number analyzed (Participants) | 84 | 75 | 77
participants | 2 | 5 | 6

2. Primary Outcome: Percentage of Heavy Drinking Days (PHDD) in the Last 4 Weeks of Treatment
Description: A heavy drinking day is defined as >= 5 standard drinking units for men and >= 4 standard drinking units for women. We calculated the PHDD used the intent-to-treat assumption, where missing drinking data were considered as heavy drinking.
Time Frame: Week 15 - 18 of the 18-week medication treatment
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
Number analyzed (Participants) | 84 | 75 | 77
percentage of heavy drinking days | 62.8 (45.4) | 65.1 (44) | 59.3 (47.3)

3. Secondary Outcome: Quality of Life in the Last 4 Weeks of Treatment
Description: We used the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) to measure quality of life in the last 4 weeks of treatment. Scoring involves summing the individual item scores on a 5-point scale, with higher scores indicating greater life satisfaction and enjoyment (better outcome). We report here a percent score of subscales contained within the Q-LES-Q, with higher scores indicating a better outcome. The subscales within the questionnaire have different numbers of items, resulting in different ranges of raw scores, so using a percent score, which used the following formula: (raw_score - scale_min_possible_score) / (scale_max_possible_score - scale_min_possible_score), helped normalize such differences, improving interpretation using the same range (i.e., 0 - 100) between subscales.
Time Frame: Week 15 - 18 of the 18-week medication treatment
Measure: Mean (Standard Deviation); unit: percent score on a scale
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
Number analyzed (Participants) | 84 | 75 | 77
percent score on a scale
  Coursework | 40.2 (6.9) | 37.1 (10.3) | 35.4 (14.4)
  General Activities | 57.7 (8.7) | 54.2 (10.7) | 57.9 (8.6)
  Household Duties | 43.6 (5.1) | 42 (7.2) | 41.6 (8.7)
  Physical Health | 25.2 (3.7) | 24.1 (4.9) | 23.4 (5.5)
  Social Relations | 51.7 (8.4) | 50.4 (10.3) | 50.8 (11.7)
  Subjective Feelings | 45.3 (6.7) | 43.6 (8.9) | 44.5 (10)
  Work | 59.2 (8.5) | 58 (10.2) | 58.9 (11.8)

4. Secondary Outcome: Craving for Alcohol and Cigarettes in the Last 4 Weeks of Treatment
Description: We used the Visual Analog Scales (VAS) to assess the craving levels for alcohol and cigarettes, respectively. VAS uses a 100 millimeter line, where 0 mm = no craving (minimum value) and 100 mm = strongest craving ever (maximum value). Participants are asked to make a mark on the line that best represents their current level of craving. Research staff then measure the distance in millimeters from the "No Craving" anchor (0 mm) to the participant's mark, which is their score. A higher score is equal to higher craving (worse outcome). Mean scores of the last 4 weeks of treatment are reported.
Time Frame: Week 15 - 18 of the 18-week medication treatment
Measure: Mean (Standard Deviation); unit: score on VAS scale
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
Number analyzed (Participants) | 84 | 75 | 77
score on VAS scale
  Craving for alcohol | 12.3 (13.9) | 18.4 (20.2) | 14.3 (14.8)
  Craving for cigarettes | 17.4 (18) | 24.6 (23.3) | 18.2 (17.8)

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected at all study visits (18 weeks), plus 30-day follow-up.
Description: Adverse events reporting followed the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 (US Department of Health and Human Services, 2017).
Arm/Group | Placebo | Low-Dose Topiramate | High-Dose Topiramate
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/75 | 0/77
Serious Adverse Events (participants affected / at risk) | 8/84 | 7/75 | 7/77
Other Adverse Events (participants affected / at risk) | 63/84 | 59/75 | 63/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Low-Dose Topiramate (N=75) | High-Dose Topiramate (N=77)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Allergic Reaction (Immune system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Concentration Impairment (Nervous system disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0
Drug Withdrawal (Psychiatric disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Neoplasms Benign, Malignant And Unspecified Incl Cysts And Polyps - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 2 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Low-Dose Topiramate (N=75) | High-Dose Topiramate (N=77)
Abdominal Pain (Gastrointestinal disorders) | 4 | 2 | 0
Agitation (Psychiatric disorders) | 8 | 8 | 7
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1
Alcohol Intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Amnesia (Psychiatric disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 12 | 11 | 9
Anal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 11 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4
Bladder Infection (Infections and infestations) | 0 | 0 | 1
Blurred Vision (Eye disorders) | 4 | 6 | 5
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Chest Pain - Cardiac (Cardiac disorders) | 4 | 2 | 3
Concentration Impairment (Nervous system disorders) | 14 | 13 | 19
Confusion (Psychiatric disorders) | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Creatinine Increased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 13 | 14 | 15
Diarrhea (Gastrointestinal disorders) | 7 | 10 | 7
Dizziness (Nervous system disorders) | 6 | 8 | 8
Drug Withdrawal (Psychiatric disorders) | 1 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 3 | 7 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 6 | 15 | 20
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1
Dysphasia (Nervous system disorders) | 0 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Edema - Face (General disorders) | 0 | 1 | 0
Edema - Limbs (General disorders) | 3 | 2 | 2
Edema - Trunk (General disorders) | 2 | 0 | 1
Ejaculation Disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 2 | 3
Eye Disorders - Other (Eye disorders) | 1 | 1 | 0
Eye Pain (Eye disorders) | 0 | 3 | 1
Fatigue (General disorders) | 16 | 13 | 19
Fever (General disorders) | 4 | 1 | 2
Flashing Lights (Eye disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0
Floaters (Eye disorders) | 0 | 1 | 1
Flu Like Symptoms (General disorders) | 7 | 4 | 11
Gait Disturbance (General disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophageal Reflux Disorder (Gastrointestinal disorders) | 1 | 3 | 1
Ggt Increased (Investigations) | 1 | 1 | 0
Gingival Pain (Metabolism and nutrition disorders) | 1 | 3 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Gum Infection (Infections and infestations) | 0 | 1 | 1
Hallucinations (Psychiatric disorders) | 2 | 0 | 2
Headache (Nervous system disorders) | 14 | 9 | 17
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1 | 2
Hemoglobin Increased (Investigations) | 1 | 0 | 0
Hyperacusis (Nervous system disorders) | 2 | 1 | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 3
Hyperosmia (Nervous system disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 6 | 5 | 9
Injury, Poisoning And Procedural Complications - Other (Injury, poisoning and procedural complications) | 7 | 10 | 7
Insomnia (Psychiatric disorders) | 20 | 20 | 13
Investigations - Other (Investigations) | 1 | 1 | 2
Irregular Menstruation (Reproductive system and breast disorders) | 1 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 7 | 9
Laryngitis (Infections and infestations) | 0 | 0 | 1
Libido Decreased (Psychiatric disorders) | 2 | 2 | 2
Libido Increased (Psychiatric disorders) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 1 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 4 | 3
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 1
Mood Alteration (Psychiatric disorders) | 3 | 0 | 1
Muscle Weakness - Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3
Nausea (Gastrointestinal disorders) | 11 | 13 | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neoplasms Benign, Malignant And Unspecified Incl Cysts And Polyps - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0
Otitis Externa (Infections and infestations) | 0 | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 9 | 5
Paresthesias (Nervous system disorders) | 10 | 21 | 38
Periorbital Edema (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 3 | 0 | 4
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Pregnancy, Puerperium And Perinatal Conditions - Other (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7 | 11
Psychiatric Disorders - Other (Psychiatric disorders) | 0 | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 0 | 1
Radiculopathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rash - Pustular (Infections and infestations) | 1 | 0 | 0
Scleral Disorder (Eye disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 8 | 7 | 10
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Speech Disorder (Nervous system disorders) | 2 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 2 | 0
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 3
Tooth Infection (Infections and infestations) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 6 | 0 | 3
Tremor (Nervous system disorders) | 0 | 3 | 0
Upper Respiratory Infection (Infections and infestations) | 11 | 6 | 11
Urinary Frequency (Renal and urinary disorders) | 3 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Urine Discoloration (Renal and urinary disorders) | 1 | 3 | 2
Urine Output Decreased (Investigations) | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Infection (Infections and infestations) | 1 | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 6 | 4
Watering Eyes (Eye disorders) | 1 | 0 | 0
Weight Gain (Investigations) | 2 | 1 | 1
Weight Loss (Investigations) | 2 | 4 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
White Blood Cell Decreased (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT01182766/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT01182766/ICF_001.pdf